CLINICAL TRIAL: NCT06881680
Title: Effects of Virtual Reality Features on Upper Limb Motor Function in Post-stroke Patients
Brief Title: Virtual Reality's Impact on Upper Limb Function in Post-stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYLL-202411-013
Record Dates: First submitted 2025-03-04; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; virtual reality (VR); body representation; upper limb dysfunction
MeSH Terms: conditions — Stroke | interventions — Smart Glasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immersive and Interactive VR group (Experimental): The design of this group combines rich immersive VR scenes and specific interactive tasks. Specifically, there were two VR scenes: (1) Natural scenery: The subjects were on a quiet forest path, surrounded by tall trees, birdsong, and the sound of gurgling water. In this scene, the program sets the virtual hand on the hemiplegic side to perform the task of grasping the sphericalfruit on the tree. Each time the fruit is grasped for 3 seconds, and then released for 3 seconds; (2) City park: The subject was located in a city park surrounded by the sounds of children playing and the background sounds of the natural environment. In this scenario, the program sets the virtual hand on the hemiplegic side to carry out the task of grasping a ping-pong ball in the park, holding it for 3 seconds at a time and then releasing it for 3 seconds. To improve the actual participation, a real object the same as the virtual object will be provided in the real world, and subjects will be instructed to use
  Interventions: Device: virtual reality (VR) head mounted display
- Interactive VR group (Active Comparator): The VR scene in this group focuses on basic motor interaction, and the virtual background is the same as the control group. The program will set the virtual hand on the hemiplegic side to complete specific interaction tasks, such as grasping the virtual ball, holding the virtual ball for 3 seconds each time, and then releasing it for 3 seconds. At the same time, a real sphere of the same size and color as the virtual ball will be provided in the real world, and the subject will be instructed to perform the same movement simultaneously as much as possible with the real hand on the hemiplegic side.
  Interventions: Device: virtual reality (VR) head mounted display
- Control group (Active Comparator): subjects were asked to wear an HTC Vive HMD and enter a simple virtual testing environment. The environment has no complex narrative or visual effects, nor does it emphasize specific interaction tasks. It only includes a realistic virtual hand model of the hemiplegic side and the same virtual background as the real experiment, both are presented from a first-person perspective. The program will set the virtual hand on the hemiplegic side to perform simple and repetitive grasping movements. Each fist hold lasts for 3 seconds and then releases for 3 seconds. At the same time, the subject will be instructed to perform the same movement simultaneously with the real hand on the hemiplegic side as much as possible.
  Interventions: Device: virtual reality (VR) head mounted display

INTERVENTIONS:
Device: virtual reality (VR) head mounted display — This group of subjects received immersive and interactive VR training, which combined rich immersive VR scenes with specific interactive tasks, including two VR scenes. Task selection was based on the subjects' upper limb functional performance, and experienced therapists provided guidance and monitoring, and adjusted the tasks when necessary.

SUMMARY:
Stroke rank second among the top causes of death, affecting millions of people in the worldwide. Approximately 70-80% survivors of stroke could experience various levels of upper limb motor impairments, which seriously affects the activities of daily life and cause serious physical and mental burden to patients and their families. As bottleneck effect in traditional rehabilitation techniques become apparent, a number of emerging technologies are being used in rehabilitation treatment in an attempt to break down this barrier.Studies have shown that virtual reality (VR) training can effectively promote the remodeling of the central nervous system and has become an important research direction for motor function rehabilitation.However, most current studies still focus on evaluating the overall intervention effect of VR, with little examination of its intrinsic properties and a lack of exploration of the sense of ownership (SOO) and agency (SOA).

Hence, this study conducted different VR interventions on stroke patients to evaluate the effects of the intrinsic properties of VR and the body illusion it produces on the rehabilitation of their upper limb motor function.

This study is a single-blind randomized controlled trial. A total of 120 participants will be enrolled and divided into a control group, an interactive VR group, and an immersive and interactive VR group. All groups will be tested on the virtual hand illusion before the intervention. The intervention will last for a fortnight, four times a week for one hour each time. Assessment will be conducted before the intervention, at the end of the intervention, and at week 6 for follow-up. The primary outcome measure is the "Fugl-Meyer Assessment of the Upper Extremity (FMA-UE)". The secondary outcome measures are "SOO questionnaire", "proprioceptive drift scale", "action research arm test (ARAT)", "NIH stroke scale (NIHSS)", "mini mental state examination (MMSE)", "electromyography (EMG)", "electroencephalography (EEG)" and "functional Magnetic Resonance Imaging (fMRI)".

ELIGIBILITY:
Inclusion Criteria:

* First episode of stroke, hemorrhagic or ischemic, confirmed by computed tomography or magnetic resonance imaging of the brain;
* Age 40-80 years, either male or female;
* 3-12 months since stroke occurrence;
* Mild-to-moderate or moderate-to-severe upper extremity impairment, with a FMA-UE score between 16 and 53;
* Basic ability to communicate and comprehend the research instructions, with a score of 21 and above on the MMSE scale;
* Agreement to participate in the study, with an informed consent form duly signed by the patient or a family member.

Exclusion Criteria:

* The presence of ferromagnetic metals implanted in the body;
* Visual or hearing deficits;
* Unstable medical conditions;
* History of receiving similar VR training in the past;
* A history of myasthenia gravis, multiple sclerosis, muscular dystrophy, or other diseases that may cause upper limb movement disorders.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Upper Extremity Scale (FAM-UE) | There were 3 time points for evaluation: before intervention, on the day of intervention end, 4 weeks after intervention end
  The Fugl-Meyer Assessment of the Upper Extremity (FMA-UE) covers all aspects of upper limb function, such as movement, coordination, and reflex actions of the shoulder, elbow, forearm, wrist, and hand, with a total of 33 assessment items. Patients were assessed according to a specific scale with a total score of 66, with higher scores indicating better recovery of upper limb function.

SECONDARY OUTCOMES:
Sense of ownership questionnaire | There were 3 time points for evaluation: before intervention, on the day of intervention end, 4 weeks after intervention end
  The sense of ownership (SOO) questionnair investigates a number of aspects including sense of body ownership, sense of position in the real or virtual hand, haptic experience, body similarity, and body transformation. Scores are allocated on a 7-point Likert scale, from "Strongly disagree (-3 points)" to "Strongly agree (3 points)", depending on how much the patient agrees with each statement. The mean score of all questions is calculated as the final SOO questionnaire score, and the higher the score, the stronger the SOO.
Proprioceptive drift scale | There were 3 time points for evaluation: before intervention, on the day of intervention end, 4 weeks after intervention end
  We asked patients to report where they thought their affected hand was by pointing with their other hand or describing it verbally and compared this with the position of the affected hand they initially felt to calculate the offset distance, thereby measuring the degree of proprioceptive error.
Action Research Arm Test | There were 3 time points for evaluation: before intervention, on the day of intervention end, 4 weeks after intervention end
  The Action Research Arm Test (ARAT) consists of 19 evaluated tasks bifurcated into four subscales: grasping, gripping, pinching, and gross motor skills. The total score ranges from 0 and 57, with higher scores representing better function.
National institutes of health stroke scale | There were 3 time points for evaluation: before intervention, on the day of intervention end, 4 weeks after intervention end
  The scale covers the level of consciousness, extraocular movements, visual fields, facial muscle function, limb strength, sensory function, coordination (ataxia), speech (aphasia), language (dysarthria), and lateralized inattention (neglect). The scoring spectrum extends from 0 to 42 points, with the higher the score, the more severe neurologic damage.
Mini-mental state examination | There were 3 time points for evaluation: before intervention, on the day of intervention end, 4 weeks after intervention end
  The Mini-Mental State Examination scale(MMSE) is mainly used to quickly assess cognitive areas such as memory, orientation, attention, calculation, language ability, and visual-spatial ability. The scale contains 30 questions with a total score range of 0-30 points. The higher the total score, the better the cognitive function. The normal threshold is divided according to the educational level (for example, those with junior high school education or above need to score ≥24 points).
Surface electromyography | There were 3 time points for evaluation: before intervention, on the day of intervention end, 4 weeks after intervention end
  Electrodes were placed on the key muscle groups of the hemiplegic upper limb according to the Surface EMG for the Non-Invasive Assessment of Muscles guidelines. In addition to the biceps and triceps brachii muscles of the upper arm, eight electrodes were placed evenly at the maximal circumference of the forearm cross-section, in which the electrodes were distributed on the centerlines of the anterior, ulnar, posterior, and radial sides of the forearm. Before placing the electrodes, the skin surface was cleaned with alcohol and the sampling rate was set to 1000 Hz. subjects were asked to perform 11 simple normative upper limb functional tasks, which were designed by Li et al. based on the FMA-UE scale . The sEMG signals were recorded during the performance of the tasks, which were repeated three times with at least 30 seconds of rest between each trial.
Electroencephalography | There were 3 time points for evaluation: before intervention, on the day of intervention end, 4 weeks after intervention end
  The subjects were seated comfortably and asked to close their eyes, wake up, relax, and be quiet for 5 minutes. The recording electrodes were placed on the scalp according to the international 10/20 system, with the Cz electrode of the head as the reference. The impedance of each channel was ensured to be below 5k Ω and the sampling frequency was 1k Hz. EEG will be used to assess changes in brain activity by analyzing the power distribution across different frequency bands (delta, theta, alpha, beta), event-related potentials (ERPs) in response to motor tasks or stimuli, and the coherence between brain regions to evaluate motor network synchronization.
functional Magnetic Resonance Imaging | There were 3 time points for evaluation: before intervention, on the day of intervention end, 4 weeks after intervention end
  The subjects were asked to remain still and provided with earplugs to alleviate discomfort from scanning noise. Functional images were acquired using an echo-planar imaging (EPI_BOLD) sequence with scanning parameters as follows: repetition time = 3000 ms, echo time = 30 ms, flip angle = 90 degrees, field of view = 220 × 220 mm, matrix size = 64 × 64, layer thickness = 3 mm layer position = 43, and a total of 240 time points being captured over a scanning period of 12 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Jinan, Shangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laver KE, Lange B, George S, Deutsch JE, Saposnik G, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2017 Nov 20;11(11):CD008349. doi: 10.1002/14651858.CD008349.pub4. PMID 29156493
- [Background] Ventura S, Tessari A, Castaldini S, Magni E, Turolla A, Banos R, Lullini G. Effectiveness of a Virtual Reality rehabilitation in stroke patients with sensory-motor and proprioception upper limb deficit: A study protocol. PLoS One. 2024 Aug 12;19(8):e0307408. doi: 10.1371/journal.pone.0307408. eCollection 2024. PMID 39133660
- [Background] Tambone R, Giachero A, Calati M, Molo MT, Burin D, Pyasik M, Cabria F, Pia L. Using Body Ownership to Modulate the Motor System in Stroke Patients. Psychol Sci. 2021 May;32(5):655-667. doi: 10.1177/0956797620975774. Epub 2021 Apr 7. PMID 33826456
- [Background] Bargeri S, Scalea S, Agosta F, Banfi G, Corbetta D, Filippi M, Sarasso E, Turolla A, Castellini G, Gianola S. Effectiveness and safety of virtual reality rehabilitation after stroke: an overview of systematic reviews. EClinicalMedicine. 2023 Sep 14;64:102220. doi: 10.1016/j.eclinm.2023.102220. eCollection 2023 Oct. PMID 37745019
- [Background] Goizueta S, Navarro MD, Calvo G, Campos G, Colomer C, Noe E, Llorens R. Touchscreen-based assessment of upper limb kinematics after stroke: Reliability, validity and sensitivity to motor impairment. J Neuroeng Rehabil. 2025 Feb 11;22(1):27. doi: 10.1186/s12984-025-01563-6. PMID 39934877
- See also: Effectiveness of Immersive Virtual Reality-Based Hand Rehabilitation Games for Improving Hand Motor Functions in Subacute Stroke Patients — https://pubmed.ncbi.nlm.nih.gov/38801680/
- See also: 360° immersive virtual reality-based mirror therapy for upper extremity function and satisfaction among stroke patients: a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/38483333/
- See also: Effects of virtual reality-based motor control training on inflammation, oxidative stress, neuroplasticity and upper limb motor function in patients with chronic stroke: a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/35016629/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-10-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT06881680/Prot_SAP_ICF_000.pdf